CLINICAL TRIAL: NCT05977439
Title: RECOVERS - Realigning Emotion and COgnition Via prEcision Regulation networkS - Phase I Study: Multimodal Computational Modeling of Cognitive Flexibility and Emotion Regulation Networks
Brief Title: RECOVERS - Realigning Emotion and COgnition Via prEcision Regulation networkS
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Columbia University (Other); University of Oklahoma (Other); Defense Advanced Research Projects Agency (U.S. Federal Agency); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 00129566
Record Dates: First submitted 2023-06-29; First posted 2023-08-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Depression - Major Depressive Disorder
Keywords: healthy volunteer; transcranial magnetic stimulation (TMS); electroencephalography (EEG); magnetic resonance imaging (MRI); functional near-infrared spectroscopy (fNIRS); cognitive behavioral therapy (CBT)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy Participants: Endorse good health with no history of mental or physical illness or implanted metal
  Interventions: Device: fMRI-EEG-TMS; Device: fNIRS-EEG-TMS
- Depressed Participants: Endorse current depression, identified via the Hamilton Depression Rating Scale (HAM-D scores ≥ 17), but no history of psychosis or mania, determined via the Quick Structured Clinical Interview for DSM-5 Disorders (SCID).
  Interventions: Device: fMRI-EEG-TMS; Device: fNIRS-EEG-TMS; Device: fNIRS-EEG-rTMS Interleaved with CBT

INTERVENTIONS:
Device: fMRI-EEG-TMS — Participants will undergo a magnetic resonance imaging (MRI) scan with combined electroencephalography (EEG), and single-pulse transcranial magnetic stimulation (TMS) while completing cognitive flexibility (CF) and emotion recognition (CR) tasks.
Device: fNIRS-EEG-TMS — Participants brain activity will be measured using functional near-infrared spectroscopy (fNIRS) with combined electroencephalography (EEG), and single-pulse transcranial magnetic stimulation (TMS) while completing cognitive flexibility (CF) and emotion recognition (CR) tasks.
Device: fNIRS-EEG-rTMS Interleaved with CBT — Participants brain activity will be measured using functional near-infrared spectroscopy (fNIRS) with combined electroencephalography (EEG), and repetitive transcranial magnetic stimulation (rTMS). rTMS will be delivered via a MagVenture MagPro100 and Cool-B65 coil. The investigators will use a standard resting motor threshold (rMT) determination to determine the TMS dose. Treatment will be delivered at 120% of the motor threshold. The accelerated paradigm will consist 6 session a day for 5-6 days. Each rTMS session will be separated by 30 minutes of Cognitive Behavioral Therapy (CBT). rTMS treatment will be delivered at an individualized left DLPFC target based on each participant's individualized scans from prior neuroimaging sessions.
  Groups: Depressed Participants

SUMMARY:
In this research study, the investigators are examining how brain activity (electrical and blood flow) changes during tests of emotional processing, attention and memory in the magnetic resonance imaging (MRI) scanner and outside the MRI using functional near-infrared spectroscopy (fNIRS). Investigators are also using non-invasive brain stimulation to probe different parts of the brain and measuring brain activity (electrical and blood flow).

Study 1

This study includes healthy participants and researchers hope this will help us develop improved brain-based treatments for emotional difficulties like depression.

Study 2

This study includes participants with depression and researchers hope this will help us develop improved brain-based treatments for emotional difficulties like depression.

DETAILED DESCRIPTION:
Investigators hypothesize that targeted neuroplastic changes induced by individually-tailored rTMS will substantially reduce clinical symptoms underlying depression, anxiety and suicidality, and in general, revolutionize non-invasive treatments of mental health disorders. Investigators hypothesize that functional coupling in cognitive flexibility (CF) and emotion regulation (ER) networks is indexed by the phase of the brain's alpha oscillations. Using a novel integrated instrument that enables simultaneous functional magnetic resonance imaging (fMRI), electroencephalography (EEG) and transcranial magnetic stimulation (TMS), investigators propose to identify individualized stimulation parameters that reflect the strongest coupling of the CF/ER networks. Investigators will also use an instrument that enables simultaneous functional near-infrared spectroscopy (fNIRS), EEG, and TMS in attempt to identify the same parameters outside the scanner. The neuromechanistic model further posits that by applying repetitive TMS (rTMS) with these individualized parameters, one can induce entrainment in brain networks that drive neuroplastic changes in CF and ER.

Study 1

This study is a proof-of-principle study in healthy control participants.

Study 2

This study is a proof-of-principle study in participants with depression.

ELIGIBILITY:
Study 1

Inclusion Criteria

* Male or female
* Age 18-65
* Endorse good health with no history of mental or physical illness or implanted metal
* English as a primary language
* Capacity to consent
* Negative urine pregnancy test if female of childbearing potential
* Willingness to adhere to the study schedule and assessments

Exclusion Criteria

* Any current psychiatric diagnosis or current Clinical Global Impression ratings of psychiatric illness > 1
* Neurodevelopmental disorders, history of CNS disease, concussion, overnight hospitalization, or other neurologic sequela, tumors, seizures, meningitis, encephalitis, or abnormal CT or MRI of the brain
* Any head trauma resulting in loss of consciousness
* Visual impairment (except the use of glasses)
* Inability to complete cognitive testing
* Active participation or plan for enrollment in clinical trial affecting the psychosocial function
* Repeated abuse or dependence upon drugs (excluding nicotine and caffeine) or taking medications including stimulants, modafinil, thyroid medication, or steroids
* Implanted devices/ferrous metal of any kind
* History of seizure or epilepsy, currently taking medications that lower seizure thresholds
* Claustrophobia or other conditions that would prevent the MRI assessment.
* Pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short term).

  o Urine Pregnancy Test: If the subject is a woman of childbearing potential and /or a man capable of fathering a child before, during, and/or after participation precautions should be taken. Examples of acceptable methods of birth control for participants involved in the study include birth control pills, patches, IUDs, condoms, sponges, diaphragm with spermicide, or avoiding sexual activity that could cause the subject to become pregnant.
* Inability to adhere to the treatment schedule

Study 2

Inclusion Criteria

* Male or female
* Age 18-65
* Endorse current depression, identified via the Hamilton Depression Rating Scale (HAM-D scores ≥ 17), but no history of psychosis or mania, determined via the Quick Structured Clinical Interview for DSM-5 Disorders (SCID).
* English as a primary language
* Capacity to consent
* Negative urine pregnancy test if female of childbearing potential
* Willingness to adhere to the study schedule and assessments

Exclusion Criteria

* Neurodevelopmental disorders, history of CNS disease, concussion, overnight hospitalization, or other neurologic sequela, tumors, seizures, meningitis, encephalitis, or abnormal CT or MRI of the brain
* Any head trauma resulting in loss of consciousness
* Visual impairment (except the use of glasses)
* Inability to complete cognitive testing
* Active participation or plan for enrollment in clinical trial affecting the psychosocial function
* Repeated abuse or dependence upon drugs (excluding nicotine and caffeine) or taking medications including stimulants, modafinil, thyroid medication, or steroids
* Implanted devices/ferrous metal of any kind
* History of seizure or epilepsy, currently taking medications that lower seizure thresholds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are healthy and depressed volunteers from the community.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in reaction time (RT) tasks - Incongruent Stimuli | Day 1, Day 2, Day 3
  Tasks will be used to see differences between incongruent emotional stimuli.
Change in reaction time (RT) tasks - Congruent Stimuli | Day 1, Day 2, Day 3
  Tasks will be used to see differences between congruent emotional stimuli.
Change in reaction time (RT) tasks and accuracy - Incongruent Stimuli | Day 1, Day 2, Day 3
  Tasks will be used to see differences between incongruent emotional stimuli.
Change in reaction time (RT) tasks and accuracy - Congruent Stimuli | Day 1, Day 2, Day 3
  Tasks will be used to see differences between congruent emotional stimuli.
Clinical Improvement | Day 13, Day 18
  25% reduction in Hamilton Score (HAMD) as a meaningful treatment response.
Clinical Improvement | Day 13, Day 18
  25% reduction in Passive and Active Suicidal Ideation Scale (PASIS) as a meaningful treatment response.
Clinical Improvement | Day 13, Day 18
  25% reduction in Patient Health Questionnaire (PHQ-9) as a meaningful treatment response.
Clinical Improvement | Day 13, Day 18
  25% reduction in Generalized Anxiety Disorder -7 Questionnaire (GAD7) as a meaningful treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McTeague, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univeristy of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No